CLINICAL TRIAL: NCT00939731
Title: A Phase I Relative Bioavailability Study To Compare The Powder-In-Capsule And Immediate Release Tablet Of PF-02341066 In Healthy Volunteers
Brief Title: Relative Drug Exposures Of Two Formulations of PF-02341066
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A8081008
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2011-10-18 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: bioavailability, capsule, tablet, healthy volunteer
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PIC (Experimental)
  Interventions: Drug: PF-02341066
- IRT (Experimental)
  Interventions: Drug: PF-02341066

INTERVENTIONS:
Drug: PF-02341066 — A 250-mg single dose of PF-02341066 administered as 1 x 50-mg Powder-in-Capsule and 2 x 100-mg Powder-in-Capsules
  Arms: PIC
Drug: PF-02341066 — A 250-mg single dose of PF-02341066 administered as 1 x 50-mg Immediate Release Tablet and 2 x 100-mg Immediate Release Tablets
  Arms: IRT

SUMMARY:
The study will be an open-label, randomized, 2-period, 2-treatment, 2-sequence, cross-over, single-dose study employing administration of two PF-02341066 formulations in the fasted state to healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non-childbearing potential subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram(ECG) and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* Pregnant or nursing females; females of childbearing potential, including those with tubal ligation. To be considered for enrollment, women of 45 to 55 years of age who are postmenopausal (defined as being amenorrheic for at least 2 years) must have confirmatory Follicle-stimulating hormone(FSH) test results at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081008&StudyName=Relative%20Drug%20Exposures%20Of%20Two%20Formulations%20of%20PF-02341066

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-02341066 250 mg IRT First, Then PF-02341066 250 mg PIC: Single oral dose of PF-02341066 250 mg immediate release tablet (IRT) in first intervention period; and single oral dose of PF-02341066 250 mg powder in capsule (PIC) in second intervention period. A washout period of at least 14 days was maintained between each period.
- PF-02341066 250 mg PIC First, Then PF-02341066 250 mg IRT: Single oral dose of PF-02341066 250 mg PIC in first intervention period; and single oral dose of PF-02341066 250 mg IRT in second intervention period. A washout period of at least 14 days was maintained between each period.
Period: First Intervention Period
Arm/Group | PF-02341066 250 mg IRT First, Then PF-02341066 250 mg PIC | PF-02341066 250 mg PIC First, Then PF-02341066 250 mg IRT
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | PF-02341066 250 mg IRT First, Then PF-02341066 250 mg PIC | PF-02341066 250 mg PIC First, Then PF-02341066 250 mg IRT
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | PF-02341066 250 mg IRT First, Then PF-02341066 250 mg PIC | PF-02341066 250 mg PIC First, Then PF-02341066 250 mg IRT
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive PF-02341066 250 mg IRT first and PF-02341066 250 mg PIC first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 32.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60, 72, 84 and 96 hours (hrs) post PF-02341066 dose in period 1 and additional 168 hrs post PF-02341066 dose in period 2
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- PF-02341066 250 mg PIC: Single oral dose of PF-02341066 250 mg PIC (Treatment A [Reference]) in either first intervention period or second intervention period.
- PF-02341066 250 mg IRT: Single oral dose of PF-02341066 250 mg IRT (Treatment B [Test]) in either first intervention period or second intervention period.
Arm/Group | PF-02341066 250 mg PIC | PF-02341066 250 mg IRT
Number analyzed (Participants) | 24 | 24
ng*hr/mL | 2804.5 (941.4) | 2597.3 (924.1)
Statistical Analysis 1: Comparison: PF-02341066 250 mg PIC vs PF-02341066 250 mg IRT; Natural log transformed AUClast of PF-02341066 was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 92.61, 90% CI 2-sided [84.84 to 101.09]

2. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60, 72, 84 and 96 hrs post PF-02341066 dose in period 1 and additional 168 hrs post PF-02341066 dose in period 2
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Median (Full Range); unit: hr
Arm/Group | PF-02341066 250 mg PIC | PF-02341066 250 mg IRT
Number analyzed (Participants) | 24 | 24
hr | 6.00 [2.00 to 8.00] | 6.00 [2.00 to 8.00]

3. Secondary Outcome: Plasma Decay Half Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-02341066 250 mg PIC | PF-02341066 250 mg IRT
Number analyzed (Participants) | 24 | 24
hr | 29.48 (4.62) | 29.10 (4.66)

4. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0 - ∞])
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-02341066 250 mg PIC | PF-02341066 250 mg IRT
Number analyzed (Participants) | 24 | 24
ng*hr/mL | 2945.5 (955.2) | 2722.5 (939.2)
Statistical Analysis 1: Comparison: PF-02341066 250 mg PIC vs PF-02341066 250 mg IRT; Natural log transformed AUC (0-∞) of PF-02341066 was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 92.43, 90% CI 2-sided [84.86 to 100.68]

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02341066 250 mg PIC | PF-02341066 250 mg IRT
Number analyzed (Participants) | 24 | 24
ng/mL | 113.35 (34.22) | 112.11 (34.87)
Statistical Analysis 1: Comparison: PF-02341066 250 mg PIC vs PF-02341066 250 mg IRT; Natural log transformed Cmax of PF-02341066 was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CI for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 98.91, 90% CI 2-sided [90.18 to 108.48]

6. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | PF-02341066 250 mg PIC | PF-02341066 250 mg IRT
Number analyzed (Participants) | 24 | 24
L/hr | 84.9 (31.6) | 91.8 (35.8)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | PF-02341066 250 mg PIC | PF-02341066 250 mg IRT
Number analyzed (Participants) | 24 | 24
L | 3566.8 (1820.5) | 3809.3 (1784.4)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-02341066 250 mg PIC | PF-02341066 250 mg IRT
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 7/24 | 8/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02341066 250 mg PIC (N=24) | PF-02341066 250 mg IRT (N=24)
Nausea (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 1 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes